CLINICAL TRIAL: NCT06904430
Title: Buckets vs Braces: Is Throw Count a Preventative Measure for Injury in Youth Throwers?
Brief Title: Buckets vs. Braces Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Kiran Athreya, Clinical Research Coordinator II, Children's Hospital of Orange County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BvB2212173
Record Dates: First submitted 2025-03-11; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Elbow Pain; Shoulder Pain
Keywords: Buckets vs. Braces
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bucket Group (Experimental): Individuals assigned to this group will limit their throw count by periodically placing the ball in a bucket over study duration
  Interventions: Other: Bucket Group
- Brace Group (Active Comparator): The participants in the brace group will be asked to wear an arm brace during baseball practice for the duration of the study
  Interventions: Device: Brace Group
- Control (No Intervention): Participants in this group will continue playing baseball with no intervention and serve as a comparison group.

INTERVENTIONS:
Other: Bucket Group — This Bucket Intervention is behavioral and studies the effect of players limiting their throw count during practice to reduce pain occurrence
  Arms: Bucket Group
Device: Brace Group — The Brace intervention studies the use of players using an elbow throwing brace during practice to reduce the occurrence of pain
  Arms: Brace Group

SUMMARY:
The purpose of this research study is to determine if there is a difference in shoulder or elbow pain between youth athletes who throw regularly without a brace, those who use a brace, and those who limit their throw count by placing the ball in a bucket during a 12-week study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 8- 12 years old
* Participation and attendance on at least 80% of practices league team
* Only participating on one baseball team for the next 12 weeks

Exclusion Criteria:

* Patients <8 or >12 years of age
* Elbow pain at the start of the season
* History of an elbow or shoulder injury, past surgeries
* Participants currently under the care of a physician for an elbow or shoulder issue
* Participants taking outside private coaching

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
To determine if there is a difference in shoulder or elbow pain between youth athletes that threw regularly without a brace, those that used a brace and those that limited their throw count by placing the ball in a bucket during a six-week study. | 12 weeks
  Shoulder and Elbow pain were assessed using the Kerlan-Jobe Orthopedic Clinic (KJOC) Shoulder and Elbow Score questionnaire. These questions are scored from 1-10 with 10 being the highest/better outcome.

SECONDARY OUTCOMES:
To identify quality of life/patient and family satisfaction with the use of limiting throw count | 12 weeks
  Participants and Families filled outcome questionnaires at baseline, midpoints, and endpoint of study responding to their satisfaction of the study and group assignments using yes/no questions, with 'yes' being the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pediatric Orthopedic Surgeon, Principal Investigator — Children's Hospital of Orange County
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States